CLINICAL TRIAL: NCT06983262
Title: Comparative Evaluation of Milled Polyether Ether Ketone (PEEK) Stent Placement and Lip Repositioning Surgery on the Treatment of Gummy Smile (A Randomized Controlled Clinical Trial)
Brief Title: Comparative Evaluation of Milled Polyether Ether Ketone (PEEK) Stent Placement and Lip Repositioning Surgery on the Treatment of Gummy Smile
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: taher helmy ismail metwaly (Other)
Responsible Party: Sponsor-Investigator, taher helmy ismail metwaly, MSc. Candidate in Periodontology, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1/3-2024
Record Dates: First submitted 2025-03-04; First posted 2025-05-21 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Gummy Smile

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VISTA and Milled PEEK stent (Experimental)
  Interventions: Other: Milled PEEK Stent
- Lip repositioning surgery (Active Comparator)
  Interventions: Procedure: Lip repositioning surgery

INTERVENTIONS:
Other: Milled PEEK Stent — A CBCT will be performed to assess the anatomy of the subnasal area and plan the position, size, shape and thickness of the PEEK Stent. These data will be transferred to a 3D planning software to generate a digital model. Eventually, the PEEK stents will be milled in a milling machine and sterilized in ethylene oxide before the surgery. Local anesthesia will be administered into the vestibular mucosa along the extension of the anterior maxilla. VISTA technique begins with a vestibular access incision in the midline frenum and 2 bilateral incisions at premolar area. A periosteal elevator will be introduced through the incision and inserted between the bone and periosteum to elevate the tissue, creating a subperiosteal tunnel, extending distally based on the dynamic of the smile. The PEEK stent will be in one piece. They will be placed onto the bone and stabilized with 2 bone graft screw for each side. The midline incision and the lateral incisions will be sutured primarily.
  Arms: VISTA and Milled PEEK stent
Procedure: Lip repositioning surgery — Profound anaesthesia will be achieved. A marking pencil§ will be used to outline the apical, coronal, and lateral boundaries of the elliptical incision. The coronal boundary will be at the mucogingival junction and will be used as a reference point to mark the apical boundary at two times the amount of gingival display. The coronal and apical incisions will be parallel to each other, and the apical incision gradually angled downward to meet the coronal incision. A partial thickness dissection will be made. The epithelium will be excised, exposing the underlying connective tissue. The mucosal flap will be advanced and sutured at the mucogingival junction.
  Arms: Lip repositioning surgery

SUMMARY:
The objective of this study is to compare between a Polyether ether ketone (PEEK) stent - and standard lip repositioning technique for management of gummy smile

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy individuals
* Chiefs complain gummy smile
* Gummy smile due to short hypermobile upper lip
* Gingival Display not more than 5 mm

Exclusion Criteria:

* Pregnancy
* Lactation
* History of smoking more than 10 cigarettes per day
* Systemic conditions or intake of medications that could affect soft and hard tissue healing
* Use of orthodontic appliances
* Gingival display above 5mm

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2024-02-14 (Actual); Primary Completion 2025-04-10 (Actual); Study Completion 2025-04-10 (Actual)

PRIMARY OUTCOMES:
Postoperative pain assessment | up to one week
  Postoperative pain will be evaluated at first and seventh day using numeric rating scale (NRS). Patient will rate his pain on a scale from 0 to 10, with 0 indicating no pain and 10 reflecting the worst possible pain.
  * 0 = no pain
  * 1-3 = mild pain
  * 4-6 = moderate pain
  * 7-10 = severe pain
Facial Edema (Swelling) | up to one week
  Postoperative edema was measured with a flexible tape measure by calculating the distance between several facial landmarks and comparing them to preoperative values.
Healing Quality | up to 3 weeks
  Measured according to Landry's Healing Index which records healing on basis of tissue colour, bleeding, ulceration, granulation tissue and epithelisation.
  Scores range from 1 (Very poor) to 5 (excellent)
Gingival display | up to 6 months
  Distance from gingival margin to lower border of upper lip vermilion border will be measured

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt